| Official Title: | Lifestyle Behavior Weight Loss<br>Intervention |
|-----------------|------------------------------------------------|
| NCT Number: | NCT04649047 |
| Document Name: | Study Protocol and Statistical Analysis Plan |
| Document Date: | November 18, 2022 |

#### Research Protocol

Weight Loss Intervention for Mothers with Young Children

## I. Objectives

- 1. Assess intervention fidelity (dose, delivery, receipt) and acceptability by the study participants
- 2. Investigate potential intervention impact on the primary (body weight) and secondary outcomes (pants size)
- 3. Explore potential intervention impact on lifestyle behaviors (diet and physical activity)
- 4. Explore potential intervention impact on motivation (autonomous motivation, self-efficacy, social support), emotion (emotion control, stress), and cognition (impulsivity).
- 5. Assess cost of different recruitment approaches

## II. Background and Rationale

Low-Income Overweight or Obese Mothers of Young Children: Our Priority Population. In the U.S., nearly 50% of low-income women aged 20-40 years are at high risk for type 2 diabetes, because they live in poverty and are overweight or obese (body mass index [BMI]  $\geq$  25.0 kg/m²).<sup>1-4</sup> One-year postpartum, low-income women have over twice the risk (68-75%) for significant weight retention ( $\geq$  10 lbs) compared to higher-income women (32%).<sup>5</sup> Significant postpartum weight retention is a strong predictor for lifelong obesity<sup>6</sup> and adverse maternal and birth outcomes, such as gestational diabetes and macrosomia<sup>7-13</sup> during subsequent pregnancies. Weight gain of  $\geq$  11 lbs during young adulthood increases risk for obesity-related conditions including type 2 diabetes,<sup>14</sup> which can be delayed and reduced by weight loss.<sup>15</sup>

**Current Lifestyle Weight Loss Intervention Studies**. Two recent meta-analyses <sup>16,17</sup> and an individual effectiveness intervention study <sup>18</sup> have shown that healthy lifestyle behaviors (healthy eating, PA) promote postpartum weight loss, including for low-income, overweight or obese women. <sup>18</sup> Despite the promise of the existing research, most prior studies have had relatively *small sample sizes*, mainly due to limitations for enrolling women within one year postpartum <sup>16,17</sup> -- high infant care demands prevent women from participating in intervention studies. <sup>16</sup> This is a missed opportunity to have broader impact on the obesity epidemic <sup>19</sup> and pregnancy-related maternal outcomes, because 40-50% of obese women gain ≥ 2 BMI units between pregnancies. <sup>20</sup> Also, prior studies *paid little or no attention to mechanisms* of motivation (autonomous motivation, self-efficacy, social support), emotion (emotion control, stress), and cognition (executive function), all of which play important roles in healthy lifestyle behaviors and resulting positive health outcomes. <sup>21-30</sup> Finally, previous lifestyle interventions have involved costly staff involvement that would be *difficult or impossible to scale up and maintain in clinical practice*. <sup>31</sup> The previous research suggests that progress is possible but fails to provide clinically-feasible and scalable options. *Thus, there is an urgent need to test scientifically rigorous, novel intervention programs, like the one that we proposed, for achieving weight loss in the priority population that could also potentially address feasibility limitations of prior work.* 

Scientific Premise. Previous research strength. Lifestyle interventions can promote weight loss. Previous research limitations. (1) The proposed priority population has been significantly underrepresented in prior lifestyle weight loss intervention studies. (2) Prior lifestyle interventions in overweight or obese mothers have suffered from threats to internal validity and have not specifically addressed motivation, emotion, and cognition (especially executive function), all of which are critical for promoting and maintaining healthy lifestyle behaviors and health outcomes. (3) There has been little evidence that any of the potentially efficacious strategies researched previously were even possible under real-world conditions. The proposed small pilot study builds on strength and effectively addresses limitations of prior research. The ultimate goal of the proposed study is to create a more feasible and scalable intervention that can be easily implemented and sustained in real-world settings. We propose to assess intervention fidelity and acceptability; we also investigate the potential utility of a web-based intervention in which participants identify their motivation for making positive behavior change, weekly goals, and means of attaining those goals, supplemented by periodic individual phone calls. Moreover, we will assess cost of different recruitment approaches. Significance. The

proposed study will add scientific knowledge on intervention implementation in a hard-to-reach population at high risk for type 2 diabetes.

## **Conceptual Framework**

Figure 1. Study Conceptual Framework



The proposed lifestyle weight loss intervention study will be the first to jointly apply future time perspective and Self-Determination Theory concepts (motivation [autonomous motivation, self-efficacy, social support], emotion (emotion control, stress), and cognition (executive function). Conceptual Framework (Figure 1). We use Future Time Perspective Theory (anticipation of future goals or personal experience across the past, present, and future<sup>32</sup>) as a guiding conceptual framework. Future time perspective drives motivation and behavior in everyday life.<sup>33</sup> Future Time Perspective Theory concepts include motivation,<sup>34</sup> emotion,<sup>33</sup> and cognition.<sup>35</sup> Implementation of future time perspective has focused on episodic future thinking.<sup>35</sup> We also apply key concepts from Self-Determination Theory: Autonomous motivation, competence (self-efficacy), and relatedness (social support), all of which foster motivation and activity engagement.<sup>36</sup> Self-Determination Theory -based interventions have effectively promoted and maintained healthy eating, <sup>22,37</sup> physical activity, <sup>38</sup> weight loss, <sup>23,39-41</sup> goal progress, <sup>42</sup> and intervention adherence. <sup>39</sup> Our **preliminary work** with the proposed priority population supports the study conceptual framework. A lifestyle intervention including stress management can effectively reduce stress<sup>43</sup> and fat intake.<sup>44</sup> Stress was positively associated with fat intake.<sup>45</sup> Self-efficacy and social support buffer stress<sup>46</sup> and dietary intake<sup>47,48</sup> Autonomous motivation and self-efficacy mediated the association between a lifestyle intervention and fat intake. 49 Self-efficacy mediated the association between a lifestyle intervention and stress.<sup>47</sup> Using an ActiGraph accelerometer (ActiGraph) to measure physical activity in the proposed population.<sup>50</sup> we found that 33.3% met physical activity recommendations (≥ 150 min/week moderate physical activity), 23.9% had some but were below the recommendations, and 42.8% had no physical activity. The proposed Goal-oriented EFT (GoEFT) intervention has two unique components that differentiate it from our own and other previous research: weekly self-directed and interactive web site (web) and individual counseling via Zoom. The vivid imagination (visualization, episodic future thinking) of goal-relevant future events in the individual's life<sup>51</sup> is specifically designed to improve motivation (autonomous motivation, self-efficacy, social support), emotion (emotion control, stress), and cognition (executive function), all of which promote success in achieving goals for healthy lifestyle behaviors. Key lifestyle behaviors include dietary intake (fewer calories, less fat and sugary drinks, and more fruit and vegetables) and physical activity (increase light-to-moderate physical activity). The proposed light-to-moderate physical activity is a realistic goal for the priority population and is consistent with public health recommendations that even modest increases in daily physical activity can yield measurable health benefits. 52-56 The primary outcome is weight loss (body weight) and the secondary outcome is waist circumference -- stronger predictors of obesity-related chronic conditions than BMI. 57-62

Connecting Episodic Future Thinking to the Proposed Mechanisms. Goal-oriented episodic future thinking<sup>29</sup> is a promising approach to improve motivation, emotion, and cognition (the proposed mechanisms connecting the intervention to the targeted lifestyle behaviors and health outcomes). Neuroimaging<sup>63-66</sup> and fMRI<sup>67-69</sup> studies have shown that episodic future thinking activates the common core network of brain regions associated with executive function during daily activity and brain regions associated with emotion regulation, decision-making, and memory. Influences on motivation: autonomous motivation, self-efficacy, and social support. Autonomous motivation -- will to engage in a behavior because of personal value, interest, or choice -- is important for achieving one's goals.<sup>36</sup> Self-efficacy refers to beliefs that one can successfully undertake an action.<sup>70</sup> Social support means receipt of various types of support, such as help from friends, family members, or others. 71 Episodic future thinking increases motivation by facilitating the link between goals and actions and by enhancing the subjective likelihood and/or value of a goal.<sup>72</sup> **Influences on** emotion: emotion control and stress. Emotion control, one's ability to manage emotional reactions using appropriate strategies, is associated with ability to cope with stress. 73 Episodic future thinking improves emotion. 67,74-76 because it activates brain regions associated with emotion regulation. 67-69 **Influences on** cognition (executive function). Executive function enables individuals to coordinate thoughts, actions, and emotions<sup>77</sup> to achieve healthy lifestyle behaviors<sup>30,78</sup> and positive health outcomes.<sup>30,77</sup> Executive function includes inhibitory control (important for EC and resisting temptation to overeat and over-react<sup>77</sup>), memory, reasoning, problem-solving, and planning. The Executive function enables individuals to take goal-directed action.<sup>78</sup> Episodic future thinking, especially goal-oriented episodic future thinking, <sup>29</sup> effectively increases inhibitory control including in overweight or obese women. <sup>28,79-81</sup> Such episodic future thinking consequences enable reduced energy intake<sup>28,29,80,82</sup> promoting weight loss<sup>83</sup> by shifting the time perspective of decision making<sup>84</sup> and activating brain areas associated with prospection.<sup>85</sup> Also, episodic future thinking fosters more relevant steps in problem solving, 86 detailed steps to attain a goal, 72 and prospective memory. 87 Finally, episodic future thinking increases reasoning, problem-solving, and planning. 67,72,86,88,89 Thus, there are many reasons to expect goal-oriented episodic future thinking to impact the proposed mechanisms.

Connecting Proposed Mechanisms to Each Other and to Lifestyle Behaviors and Health Outcomes. Motivation and emotion are inter-related components of self-regulation that enable individuals to adhere to a healthy lifestyle and achieve positive health outcomes. 90 **Motivation**. Increased autonomous motivation, self-efficacy, and social support are strongly associated with reducing stress in overweight or obese women<sup>46,47,91</sup> and with promoting cognitive performance<sup>92</sup> (e.g., problem solving<sup>93</sup>) and a healthy lifestyle.<sup>21</sup>-<sup>25,47,48,94</sup> Also, autonomous motivation predicts successful goal pursuit<sup>32,95</sup> and promotes weight management. 24,40,96,97 Emotion influences cognition. 98 Stress negatively affects diet (increased intake of highfat, sugary, energy-dense foods, leading to weight gain<sup>27</sup>) and physical activity.<sup>26</sup> Higher levels of stress are associated with lower levels of inhibitory control<sup>27</sup> and interfere with cognitive performance, <sup>99</sup> but reducing stress improves executive function. 100 Cognition (executive function). Low levels of inhibitory control have been associated with increased energy intake in overweight or obese women, 79 but high levels of inhibitory control have been associated with reduced consumption of total calories, percent calories from fat, 28,29 and snacking and food intake<sup>80,82</sup> in women. Executive function also predicts moderate-to-vigorous PA,<sup>30</sup> maintenance of PA,<sup>101</sup> and weight loss.<sup>30</sup> Executive function deficits are more likely in overweight or obese than normal-weight women 102-105 and can be improved through training and practice. 100 Thus, previous research supports associations among the key mechanisms and connects those mechanisms to healthy lifestyle behaviors and to health outcomes.

The study would also be the first to apply episodic future thinking outside the lab with no in-person component (emphasizing clinical feasibility). The use of episodic future thinking is more effective for long-term motivation and planning than self-generated thought without episodic future thinking. Episodic future thinking enables individuals to generate detailed goal-relevant scene construction, 64,88,106,107 whereas self-generated thought without episodic future thinking focuses on behaviors with minimum or no scene construction. With the exception of one "internet plus in-person" four-week intervention, 33 all prior episodic future thinking studies have been conducted in lab settings where participants followed intensive and specific scripts directing them through vivid imagination of future events. Thus, the relevance and scalability of episodic future thinking for clinical practice remains speculative. Moreover, prior episodic future thinking studies have only focused on one

form of *episodic future thinking*: episodic simulation (mental representation of the future). <sup>67</sup> The proposed intervention includes episodic simulation, prediction (benefits for achieving goals), intention (identifying when and where the activity will take place), and planning (generating specific steps rather than general plans for achieving the goal done by prior research), all of which come together to support prospective cognition. <sup>109</sup> Furthermore, the study would be *the first to ask participants to vividly imagine their personal plans followed by enabling them to weekly customize the plans*. This approach supports the sense of volition and choice and fulfilling the psychological needs of the participants, which in turn promotes quality of intervention engagement and outcomes. <sup>110</sup> Finally, the study would innovate in *use of participant-generated short reminders to promote cohort retention and intervention dosage.* <sup>111</sup>

### A. Research Design

This pilot quasi experimental design study aims to (1) assess intervention fidelity (dose, delivery, receipt) and acceptability by the study participants, (2) investigate potential intervention impact on the primary (body weight) and secondary outcomes (waist circumference), (3) explore potential intervention impact on lifestyle behaviors (diet and physical activity), (4) explore potential intervention impact on motivation (autonomous motivation, self-efficacy, social support), emotion (emotion control, stress), and cognition (impulsivity), and (5) assess cost of different recruitment approaches. We will enroll 30 overweight or obese women with diverse racial and ethnic backgrounds. All measures will be assessed at baseline (T1) and immediately after the three-week intervention (T2).

### B. Sample

#### Inclusion Criteria. Self-reported

■ BMI of 25.0-45.0 kg/m² (calculated using height and weight) ■ Current enrollment in government assistant programs (for example, WIC, food stamp (SNAP), or Madicaid) ■ 6 weeks - 5 years postpartum ■ 18-45 years old ■ Fluency in speaking, reading, and writing English ■ Ownership of a smart phone with unlimited text messages and internet access ■ Committed to a three-week intervention study

## **Exclusion Criteria.** Self-reported

■ Current pregnancy or lactation ■ Plan to become pregnant during the trial ■ Type 1 or 2 diabetes ■ Untreated thyroid disease ■ Drug or alcohol abuse or dependence within last six months ■ Major psychiatric disorder (e.g., schizophrenia, bipolar) ■ History of bulimia or anorexia ■ Current taking of appetite suppressant or (antipsychotic) medications known to affect body weight ■ Current participation in a weight control or drug study ■ Current or planned participation in a commercial weight loss program ■ Previous weight loss surgery ■ Contraindications to physical activity.

**Sample size/power.** We did not perform a formal sample size calculation but based on our available funding and resources. Because of budget constraint, we think a sample size of 30 women is appropriate for this pilot, which will provide preliminary data for us to apply future NIH R01.

### C. Measurement/Instrumentation

All participants will be assessed at baseline (T1) and immediately after the three-week intervention (T2). Survey data will be collected online using password-protected security-ensured Research Electronic Data Capture (REDCap), a secure web application for building and managing online surveys and databases. Participants will receive up to \$10 for completing T1 data collection and \$20 for T2 data collection. We will contact participants to verify or clarify survey data, e.g., body weight is entered as 90 (most unlikely because we will enroll overweight or obese women) instead of 190.

**Feasibility.** We will use our tracking records to assess <u>recruitment and retention.</u> To assess <u>intervention implementation,</u> we will extract data from our study web site that will track and capture details about all activities (e.g., amount of and type of activities completed and percent of participants used type in box). We will record the attendance of individual coaching session. Participants will report their motivation and barriers preventing them from engaging in the intervention activities and evaluate the usefulness of with each episodic

future thinking intervention component. We will also use semi-structure interview questions (up to 20 minutes/an individual interview via zoom) to ask participants to evaluate the intervention. We will use website tracking data, individual coaching session, and results of zoom interview to revise the intervention contents for a future large scale intervention study (R01).

**Primary outcome**: body weight. We will collect self-reported body weight.

**Secondary outcome**: waist circumference. We will collect self-reported pants size, which is a good indicator of waist circumference.

### Lifestyle behaviors.

**Dietary fat.** The NCI brief dietary fat intake survey (16 items)<sup>112</sup> will be used to measure dietary fat intake. Participants will be asked about frequency of consuming a list of foods. **Fruit and vegetable intake**. NCI five factor screener (9 items)<sup>113</sup> will be used to measure fruit and vegetable intake. Participants will be asked about the frequency of eating fruit and vegetables. **Sugar intake**. NCI five-factor screener (4 items)<sup>114</sup> will be used to measure sugar intake. Participants will be asked about the frequency of eating foods and sweeten beverage. **Physical activity**. The International Physical Activity Questionnaire Short Form (7 items)<sup>115</sup> will be used to measure physical activity. Participants will be asked amount of time spent on physical activities.

## Concepts.

*Motivation*. *Autonomous motivation* will be measured using Treatment Self-Regulation Questionnaire (18 items) that asks why the respondent does a behavior. Self-efficacy will be measured using a 10-item survey for general self-efficacy, and a 10-item survey for healthy eating self-efficacy, and a 10-item survey for physical activity self-efficacy, that ask participants confidence in performing the specific activity. Social support measures ask mothers to report social support from their family members, friends, or other people to manage stress (6 items), eat healthier (6 items), and engage in PA (4 items). Emotion. Emotion control will be measured using the Emotion Regulation Questionnaire (10 items) that assess emotion regulatory process using reappraisal, suppression and regulating negative emotion. Stress will be measured using The Perceived Stress Scale (10 items) that measures the degree to which situations in one's life are appraised as stressful. Cognition. To measure executive function (impulsivity), we will use Barratt Impulsiveness Scale (30 items) to measure impulsivity.

### Process evaluation.

All participants will report receipt of lifestyle behavior counseling from their clinicians, midwifes and dietitians and joining other programs.

#### Recruitment cost

We will track time and effort spend on each recruitment method.

## Sent messages to participants

We will email and text participants to complete study activates. Please note the sequence listed below corresponding to the sequence listed on the file called "All Email and Text Messages."

| Activities | Email | Text | Notes |
|---|---|---|---|
| A. Enrollment Phase | | | |
| A1. Attend information session (first zoom meeting) | Yes | Yes | Up to 3 times |
| A2. Full consent to participation | Yes | No | Up to 3 times |
| A3. Attend second zoom meeting | Yes | Yes | Up to 3 times |
| B. Intervention Phase | | | |
| B1: Complete Part I intervention: | Yes | Yes | Need to send both email and text (at the same time) |
| becoming a better me | | | because of including web link—participants can |

| | | | complete via smart phone or computer internet access. Up to 3 times for each |
|---|---|---|---|
| B2. Complete Part II intervention: safe care booster | Yes | Yes | Need to send both email and text (at the same time) because of including web link. Up to 3 times for each |
| B3. Join the weekly individual coaching via zoom | Yes | Yes | Up to 3 times |
| C. Throughout the project | | | |
| C1. Fill out online survey | Yes | Yes | Need to send both email and text (at the same time) |
| | | | because of including web link. Up to 3 times for each |
| D. Notify Incentives | Yes | Yes | Up to 3 times for each |

## E. Detailed study procedures

**Recruitment and enrollment**. Participants will be recruited via four approaches: (1) FaceBook, (2) Study Search, (3) Research Match, (4) MyChart, and (5) study flyer

**FaceBook**, We will post the study flyer at FaceBook (File name: Flyer\_FaceBook Add). Potential participants who are interested in the study will contact the study office for screening.

**Study Search**. We will post the study flyer at Study Search via OSU Medical Center website (File name:Flyer\_study search). Potential participants who are interested in the study will contact the study office for screening.

**Research Match.** We will post the study flyer at Research Match website (File name: Flyer\_Research Match, which describe how participants will be identified in details). The study office will contact the potential participants who are interested in the study.

**MyChart.** We will post the study flyer at MyChart (via 'OSU BMI', File name: Flyer\_MyChart). Upon IRB approval, we will submit an "honest broker data request form" followed by working with 'OSU BMI' to identify potential participants. Once potential participants who are interested in the study are identified, 'OSU BMI' will refer these potential participants to IHIS box. The trained research staff will log into IHIS to contact the potential participants.

**Study Flyer**. We will post the study flyer in, for example, clinics, website (e.g., Craig's list, google). We will also ask organizations that agree to collaborate with us to send the study flyer via email or other social media to their clients or customers. Potential participants who are interested in the study will contact the study office for screening.

<u>Initial Contact of Potential Participants</u> regardless methods of recruitment. We will obtain verbal consent prior to screening and obtaining demographic information. Collecting demographic data will help us revise or plan for recruitment strategies for a future R01. If eligible, participants will provide up to three working telephone numbers (at least one capable of receiving text messages), email address, and physical address as contact information. We will ask if we can leave a message via phone (Yes/No). Next, the Research Staff will schedule a zoom meeting (individual information session, described below) within the five business days with the qualified participants (we will allow extension if participants indicate the time line does not work for them). Then, the trained research staff will send the full consent form to the participants for review (via email) prior to the first scheduled zoom meeting. Participants will be informed the zoom meeting will be either audio or video recorded per their preferences.

First zoom meeting (information session lead by research staff). Participants will use their personal devise, for example, computer or smartphone to join the zoom meeting, which will take up to 40 minutes. First, the trained research staff will ask participants if they have questions and answer questions accordingly. Next, they will review key summary of incentive and intervention requirements (using Zoom "share") with the participants and answer questions that they may have. Also, research staff will ask the potential participants to think through their current and anticipated responsibilities and life situations before providing electronic signature (via REDCap) for participation. After that, the research staff will obtain consent (participants providing electronic signature via REDCap) followed by showing them how to complete the online survey and requirements. Then, participants will be asked to self-generate reminders to complete data

collection activities. Finally, participants will be informed about the purpose of the second zoom meeting. They will also be informed that they must complete the online survey within three weeks of the first Zoom meeting in order to be invited to attend the second zoom meeting.

<u>Second zoom meeting (either audio or video recorded per participant preferences.</u> Participants will be enrolled. First, they will be asked to self-generate 3-5 text messages to remind them to complete the intervention activities and join brief individual coaching via Zoom. Next, they will receive a link to complete part I intervention activities, which will take up to 35 minutes to complete. Participants will use their first and last name, and birthday and own device (e.g., smart phone) to log into the intervention website and complete activities, while the research staff still on Zoom to answer women's questions if they have. After completion of the Part I intervention activities, the research staff will schedule an individual coaching session via zoom with the trained interventionist within the next two days. Participants will be informed that each coaching session will be recorded (either audio or video per their preferences). The recording will be transcribed and be analyzed to help us revise the individual coaching sessions for future studies. We will send a zoom link to participants to join the individual coaching session.

**Cohort retention.** We will apply our previously successful retention strategies. We will allow temporary lapses as needed (e.g., partial data collection at T2) or extend the time window for data collection. We will monitor the retention rate monthly and keep retention logs by asking participants over the phone about their reasons for dropout and any adjustments that could keep them in the study.

Intervention: A self-directed, web-based lifestyle behavior intervention (tailored to participants' needs). *Intervention mode.* All intervention participants will receive the weekly web-based intervention for three weeks. The intervention includes *three topics*: stress management, healthy eating, and physical activity (Figure 2). *Intervention (long-term) goals.* Participants are strongly encouraged to (1) daily manage stress and emotional reactions using positive strategies, (2) daily eat a diet low in fat and consume less sugary drinks, (3) daily eat a diet high in fruits and vegetables, and (4) walk at a brisk pace for 30 min most days a week.<sup>56</sup>

**Figure 2. Topics for the three-week intervention.** *Stress management* includes three subtopics (e.g., better ways to handle everyday life) and 13 short-term goals (e.g., have a better relationship with family). *Healthy eating* includes four subtopics (e.g., effective ways to reduce junk food intake) and 11 short-term goals (e.g., daily eat less junk food and be mindful what I eat). *Physical activity* has one subtopic and three short-term goals (e.g., being more physically active outdoors).

| | Week 1 | Week 2 | Week 3 |
|---|---|---|---|
| Weekly web (up to 40 min/week) | Stress | Healthy eating | Physical activity |
| | management | | |
| Weekly individual coaching via zoom | Х | Х | Х |
| (15 min/call, 10 calls) | | | |

Intervention development based on preliminary work. *Informal interviews with stakeholders*. We informally met with several clinicians who provided prenatal care to the target audience to inform our mode of intervention delivery. They suggested a self-directed, web-based intervention because of its easy implementation and future scalability to overcome clinicians' time constraints to providing additional information on stress management, healthy eating and physical activity to help women manage their weight. *Study one.* We conducted seven focus group discussions with overweight or obese pregnant women (N = 96) to identify their critical needs in stress management, healthy eating, and physical activity. Women reported, for example, poor relationships with significant others, feeling emotional, eating foods for comfort, and lack of motivation to be physically active. Passing this study were used to develop the pre-written short-term goals for the participants (Figure 2) because most women had challenges in goal setting. *Study two*. Below, we present lessons learned from our prior NIH-NIDDK R18 intervention study of overweight or obese women of child-bearing age<sup>124</sup> to develop the two parts of the GOEFT intervention (Figure 3). Part I. *Motivation*. Lesson learned: Personal values and interest (autonomous motivation) motivated women to make positive lifestyle

behavior changes. Many women had low commitment and confidence (self-efficacy) to implement plans/steps to achieve personal values and make positive changes. *Emotion and cognition*. Lesson learned: Realizing the importance (i.e., the potential benefits) of accomplishing personal goals and responding to open-ended questions (e.g., WHAT and WHY) helped women aware of current life situations/challenges and motived them to make positive changes. Yet, most women faced challenges in setting goals and identifying specific steps to accomplish the goals. Also, many challenges (e.g., lack of willpower, time, or energy) prevented them from implementing their plans. Including explicit planning and (HOW) material for how to overcome challenges should buttress the effectiveness of the current intervention. Part II: *Evaluation of goal progress with feedback*. Lesson learned: women were often unaware what strategies helped them accomplish their goals. They often gave up when unaware of the progress toward their goals or the benefits received from making positive changes. *Based on the conceptual framework (Figure 1) and results of the preliminary work, Drs. Chang (an expert in healthy lifestyle behavior interventions including stress management) and Wegener (Co-I, an expert in psychological emotion and cognition research) worked with five peers of the target audience to develop the* 

# Figure 3. A three-week self-directed, web-based intervention (35-40 min/week)

## Part 1 (Weekly Days 1-4: 30-35 min)

# Motivation (Autonomous motivation, self-efficacy)

-Three most important personal values, ways to commit to personal values followed by ways to boost confidence in achieving personal values

# Emotion (emotion control, stress) and Cognition (Executive function)

-The first short-term goal, WHAT (the week's goal), WHY(importance of the goal), WHEN and WHERE (the goal taking place), WHO (persons involved in the goal) and HOW (generating three steps to achieve the goal) followed by selecting the second short-term goal and repeating five Ws and H

#### Motivation (self-efficacy)

-Three daily challenges to implement the steps, three solutions to each of the chosen challenge, and benefits of overcoming chosen challenges.

Summary of part I

### Part II (Weekly Days 5-7: 5 min)

## **Evaluation of Goal Process with Feedback**

-Two short-term goals, helpful tips used to achieve the goals, benefits of achieving the goals, four long-term goals followed by personal values

Summary of part II

proposed self-directed, web-based goaloriented episodic future thinking intervention (Figure 3). After developing the draft intervention, we used feedback from several additional peers of the target audience to review and finalize the intervention.

#### Intervention

**implementation** (Figure 3). Research staff will provide the intervention web link (via text, email) and instructions on completing the weekly intervention activities online. Intervention participants will use their smart phone, first and last name, and birthday to log into the website to complete the Part I intervention activities for week one. Week one Part I activity will be completed during the second zoom meeting to increase participants interest in participation. Also, research staff will answer any questions that participants may have. The day of the week that the participants complete the Part I intervention activities will count as their weekly day one. All participants will be given the study office number to call for questions and technical problems.

Participants will use their own device to complete Part II intervention activities for week one and the additional two weeks of the intervention at convenient times and locations. We will send the web link to participants weekly via email and text with an "intervention adherence" text message reminder (generated by the participants) to log in and complete the intervention activities.

Part I (weekly days 1-4, 30-35 min/week): Motivation, emotion and cognition. *Motivation*. Participants will first be asked to visualize, then use a dropdown menu to select their responses (or type in a box) for the following: their personal values and ways to help them commit to and increase confidence in achieving their personal values. *Emotion and cognition*. First, participants will select a subtopic from the week's designated topic (Figure 2) followed by selecting a pre-written short-term goal (or typing in a box) under the chosen subtopic that meets their need for that week's focus. Then, they will visualize and describe WHAT the week's goal is, WHY it is important, WHEN, WHERE, and with WHOM it will take place, and HOW it can be

accomplished, all of which enhance prospective memory, thus enabling individuals to carry out the plan to reach the goal. 125 Related to HOW, they will be asked to view an example with three specific detailed steps to achieve their chosen goal. Step I. Use open-ended questions to ask themselves, thus to raise awareness of their current life situations/challenges (e.g., How often do I eat junk foods?). Step II. Take specific steps to overcome the challenges to achieve the chosen goal (e.g., pay attention to foods I eat and how much I eat). Step III. Record ways to reward themselves without using foods (e.g., smile and tell myself, "Wow, I am proud of myself of eating less junk food and being mindful what I eat, each time I follow through my plans"). After that, participants will visualize and describe their three steps (by typing) to accomplish the chosen goal. Next, they will repeat the same process for a second short-term goal for the week. *Motivation*. they will visualize and use the dropdown menus to select (or type in a box) (1) their three most important challenges (e.g., I don't have the willpower) in implementing their steps to accomplish each of chosen goal for the week, (2) three potential solutions to overcome each chosen challenge and (3) benefits of overcoming the challenges. Phase I concludes with a summary of the participant's motivation, emotion and cognition. Participants will be encouraged to accomplish their chosen goal within the next few days and mentally rehearse their "identified steps" two times daily because rehearsal increases effectiveness of goal-oriented episodic future thinking on the chosen goals. 126

Part II (weekly days 5-7, 5 min/week): Evaluation of goal progress with feedback. After implementing steps to achieve both chosen goals, they will log into the intervention website and use the dropdown menus to evaluate their progress on accomplishing their short-term goals, identify tips that proved helpful, recognize short- and long-term benefits of accomplishing the chosen goals, and rate progress on the four long-term intervention goals and three chosen personal values. They will receive feedback to their response for each evaluation component (e.g., short-term goal). Part II concludes with a summary of goal progress with feedback.

Individual coaching session via Zoom (15 min/call, 10 calls). Participants will receive a call within 1-2 days after they complete the Part I intervention activities. All coaching session will be either video or audio recorded (per participants' preference) with participants' permission. Participants will be informed that the recording will be transcribed and be used to refine the individual coaching session for future studies. During each call, the research will listen empathetically and use open-ended questions asking participants to visualize and describe how the week's goals fit with their personal values, thereby supporting their motivation (autonomous motivation). Next, participants will be asked to visualize and describe how they will accomplish the goal(s) – what specific steps they will take. Then, the research staff will assess the specificity of the steps and reinforce or help modify the plans (emotion and cognition). Finally, participants will be asked to visualize and describe barriers to implement plans and strategies to overcome barriers. The research staff will assist with problem solving as needed (self-efficacy). We will keep IPC attendance records. Fidelity. Dr. Chang and each research will listen to a random 25% of the audio recordings monthly and use the fidelity checklist to assess protocol adherence, strengths, and reasons for deviations.

Intervention adherence. Each week, participants will receive up to three prescheduled text reminders via their smart phone to engage in the week's intervention activities (until they complete). If women have not completed all activities after seven days, the research staff will call and ask them to complete the activities that they have missed and ask reasons for nonadherence. When a woman expresses interest in quitting some aspects of the intervention activities, we will assess barriers to adherence, brainstorm strategies to overcome barriers, and offer options to reduce intervention adherence burden. We will keep intervention adherence log.

# F. Internal Validity

**Feasibility of recruitment, retention, intervention adherence and acceptability (Aim 1)**. We already plan to track *recruitment and retention* activities. *Intervention adherence*. The web will track and capture details about all activities (e.g., number of logins and amount of and type of contents used). We will also ask intervention participants about motivation and barriers preventing them from using the web. *Acceptability*. We will assess acceptability by asking participants to evaluate the usefulness of with each intervention component,

e.g., personal values, using 5 Ws and H, and rehearsal. Lessons learned and results of this aim will be used to refine our future R01, e.g., recruitment and intervention.

**Measures (See above and File Name: Study Survey. shown above).** Self-reported data will be collected online using password-protected security-ensured Research Electronic Data Capture (REDCAP).

## G. Statistical analysis

**Statistical analysis.** We will use descriptive statistics to examine variable distributions, check for outliers, and summarize sample characteristics. **Aim 1.** We will (1) conduct content analysis to analyze recruitment, enrollment, retention and intervention adherence logs to identify successful strategies used, (2) review quality of steps generated to achieve goals (using a scoring system), and (3) perform descriptive statistics. We will also perform content analysis (for semi-structure interview questions). **Aims 2, 3, and 4. Aim 5.** We will perform descriptive analysis. We will first preform descriptive statistics. Next, we will preform mixed-effects linear modeling. **Missing data**. We will carefully examine the pattern of missing data and conduct appropriate multiple imputation if missing at random is indicated. The mixed-effects modeling allows for missing at random. If missing not at random exists, pattern mixture modeling will be used. Sensitivity analysis will evaluate the robustness of study findings without multiple imputation vs. those with imputation or from pattern-mixture modeling.

## **Zoom IRB Boilerplate:**

Zoom is a secure, user-friendly, cloud-based enterprise videoconferencing service that Ohio State University implemented in 2018. Zoom is accessible to faculty and staff at all Ohio State campuses via <a href="https://carmenzoom.osu.edu">https://carmenzoom.osu.edu</a>.

This multifaceted video and audio conferencing system supports video and audio conferencing across multiple platforms, including room systems, mobile devices, desktops and telephones.

The Zoom platform at Ohio State University has two main features: Zoom meetings and Zoom webinars.

Designed to support collaboration, Zoom meetings support up to 300 video participants. By default, any participant in a meeting can share their video and audio and utilize the chat feature to exchange messages with participants. The meeting host controls all meeting features, which include mute/unmute participants, screen sharing, recording options, video sharing, remote screen control and participant annotation. Annotation allows participants to draw and highlight on the screen share. Zoom webinar provides access for up to 300 view-only attendees and features live question-and-answer, polling, registration and post-webinar reporting.

Ohio State University Zoom offers both local recording and cloud recording and has a storage capacity of 270 days for recordings. Cloud recording includes an option to produce an audio transcript for a meeting or webinar. The transcript is saved to the cloud as a separate .vtt text file, and the host can elect to display the transcript text within the video itself, similar to a closed-caption display.

Zoom is accessed via Ohio State's single sign-on solution, which provides an environment in which users can authenticate/log in at one time to a central server and connect with web-based services. Meeting security best practices such as waiting lobby, inability to join before host, disabling of sharing for participants, and disabling annotation by participants by default have been implemented.

## III. Bibliography

- 1. Prevention CfDCa. Eligibility and enrollment in the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC)--27 states and New York City, 2007-2008. MMWR Morb Mortal Wkly Rep. 2013:62(10):189-193.
- 2. Bullard KM, Cowie CC, Lessem SE, et al. Prevalence of Diagnosed Diabetes in Adults by Diabetes Type United States, 2016. *MMWR Morb Mortal Wkly Rep.* 2018;67(12):359-361.
- 3. Hales CM, Fryar CD, Carroll MD, Freedman DS, Aoki Y, Ogden CL. Differences in Obesity Prevalence by Demographic Characteristics and Urbanization Level Among Adults in the United States, 2013-2016. *JAMA*. 2018;319(23):2419-2429.
- 4. Braveman PA, Cubbin C, Egerter S, Williams DR, Pamuk E. Socioeconomic disparities in health in the United States: what the patterns tell us. *Am J Public Health*. 2010;100 Suppl 1:S186-196.
- 5. Endres LK, Straub H, McKinney C, et al. Postpartum weight retention risk factors and relationship to obesity at 1 year. *Obstet Gynecol.* 2015;125(1):144-152.
- 6. Rooney BL, Schauberger CW. Excess pregnancy weight gain and long-term obesity: one decade later. *Obstet Gynecol.* 2002;100(2):245-252.
- 7. Doherty DA, Magann EF, Francis J, Morrison JC, Newnham JP. Pre-pregnancy body mass index and pregnancy outcomes. *Int J Gynaecol Obstet*. 2006;95(3):242-247.
- 8. Villamor E, Cnattingius S. Interpregnancy weight change and risk of adverse pregnancy outcomes: a population-based study. *Lancet*. 2006;368(9542):1164-1170.
- 9. Heslehurst N, Simpson H, Ells LJ, et al. The impact of maternal BMI status on pregnancy outcomes with immediate short-term obstetric resource implications: a meta-analysis. *Obes Rev.* 2008;9(6):635-683.
- 10. Koebnick C, Smith N, Huang K, Martinez MP, Clancy HA, Kushi LH. The prevalence of obesity and obesity-related health conditions in a large, multiethnic cohort of young adults in California. *Ann Epidemiol*. 2012;22(9):609-616.
- 11. Baeten JM, Bukusi EA, Lambe M. Pregnancy complications and outcomes among overweight and obese nulliparous women. *Am J Public Health*. 2001;91(3):436-440.
- 12. Kabali C, Werler MM. Pre-pregnant body mass index, weight gain and the risk of delivering large babies among non-diabetic mothers. *Int J Gynaecol Obstet*. 2007;97(2):100-104.
- 13. Johansson S, Villamor E, Altman M, Bonamy AK, Granath F, Cnattingius S. Maternal overweight and obesity in early pregnancy and risk of infant mortality: a population based cohort study in Sweden. *BMJ*. 2014;349:g6572.
- 14. Zheng Y, Manson JE, Yuan C, et al. Associations of Weight Gain From Early to Middle Adulthood With Major Health Outcomes Later in Life. *JAMA*. 2017;318(3):255-269.
- 15. LeBlanc ES, Patnode CD, Webber EM, Redmond N, Rushkin M, O'Connor EA. Behavioral and Pharmacotherapy Weight Loss Interventions to Prevent Obesity-Related Morbidity and Mortality in Adults: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. *JAMA*. 2018;320(11):1172-1191.
- 16. Lim S, O'Reilly S, Behrens H, Skinner T, Ellis I, Dunbar JA. Effective strategies for weight loss in post-partum women: a systematic review and meta-analysis. *Obes Rev.* 2015;16(11):972-987.
- 17. Lim S, Liang X, Hill B, Teede H, Moran LJ, O'Reilly S. A systematic review and meta-analysis of intervention characteristics in postpartum weight management using the TIDieR framework: A summary of evidence to inform implementation. *Obes Rev.* 2019;20(7):1045-1056.
- 18. Phelan S, Hagobian T, Brannen A, et al. Effect of an Internet-Based Program on Weight Loss for Low-Income Postpartum Women: A Randomized Clinical Trial. *JAMA*. 2017;317(23):2381-2391.
- 19. McKinley MC, Allen-Walker V, McGirr C, Rooney C, Woodside JV. Weight loss after pregnancy: challenges and opportunities. *Nutr Res Rev.* 2018;31(2):225-238.
- 20. Jain AP, Gavard JA, Rice JJ, Catanzaro RB, Artal R, Hopkins SA. The impact of interpregnancy weight change on birthweight in obese women. *Am J Obstet Gynecol*. 2013;208(3):205 e201-207.
- 21. Senecal C, Nouwen A, White D. Motivation and dietary self-care in adults with diabetes: are self-efficacy and autonomous self-regulation complementary or competing constructs? *Health Psychol.* 2000;19(5):452-457.
- 22. Shaikh AR, Vinokur AD, Yaroch AL, Williams GC, Resnicow K. Direct and mediated effects of two theoretically based interventions to increase consumption of fruits and vegetables in the Healthy Body Healthy Spirit trial. *Health Educ Behav.* 2011;38(5):492-501.
- 23. Silva MN, Vieira PN, Coutinho SR, et al. Using self-determination theory to promote physical activity and weight control: a randomized controlled trial in women. *J Behav Med.* 2010;33(2):110-122.

- 24. Teixeira PJ, Carraca EV, Marques MM, et al. Successful behavior change in obesity interventions in adults: a systematic review of self-regulation mediators. *BMC Med.* 2015;13:84.
- 25. Santos I, Ball K, Crawford D, Teixeira PJ. Motivation and Barriers for Leisure-Time Physical Activity in Socioeconomically Disadvantaged Women. *PLoS One.* 2016;11(1):e0147735.
- 26. Chang M, Nitzke S, Guilford E, Adair C, Hazard D. Motivators and barriers to healthful eating and physical activity among low-income overweight and obese mothers. *J Am Diet Assoc.* 2008;108(6):1023-1028.
- 27. Fields SA, Lange K, Ramos A, Thamotharan S, Rassu F. The relationship between stress and delay discounting: a meta-analytic review. *Behav Pharmacol*. 2014;25(5-6):434-444.
- 28. Daniel TO, Stanton CM, Epstein LH. The future is now: comparing the effect of episodic future thinking on impulsivity in lean and obese individuals. *Appetite*. 2013;71:120-125.
- 29. O'Donnell S., Oluyomi Daniel T., LH E. Does goal relevant episodic future thinking amplify the effect on delay discounting? *Conscious Cogn* 2017;51:10-16.
- 30. Butryn ML, Martinelli MK, Remmert JE, et al. Executive Functioning as a Predictor of Weight Loss and Physical Activity Outcomes. *Ann Behav Med.* 2019.
- 31. Garfield SA, Malozowski S, Chin MH, et al. Considerations for diabetes translational research in real-world settings. *Diabetes Care*. 2003;26(9):2670-2674.
- 32. Lens W, Paixao MP, Herrera D, Grobler A. Future time perspective as a motivational variable: Content and extension of future goals affect the quantity and quality of motivation. *Japanese Psychological Research*. 2012;54(3):321-333.
- 33. Andre L, van Vianen AEM, Peetsma TTD, Oort FJ. Motivational power of future time perspective: Meta-analyses in education, work, and health. *PLoS One*. 2018;13(1):e0190492.
- 34. Kooij D, Kanfer R, Betts M, Rudolph CW. Future time perspective: A systematic review and meta-analysis. *J Appl Psychol.* 2018;103(8):867-893.
- 35. Husman J., J.C H. Extending Future Time Perspective Theory through Episodic Future Thinking Research: A Multidisciplinary Approach to Thinking About the Future. In: Kostić A. CDe, ed. *Time Perspective*. London: Palgrave Macmillan; 2017:267-280.
- 36. Deci EL, Ryan RM. The "What" and "Why" of Goal Pursuits: Human Needs and the Self-Determination of Behavior. *Psychological Inquiry*. 2000;11(4).
- 37. Robles B, Smith LV, Ponce M, Piron J, Kuo T. The influence of gender and self-efficacy on healthy eating in a low-income urban population affected by structural changes to the food environment. *J Obes.* 2014;2014:908391.
- 38. Cramp AG, Bray SR. A prospective examination of exercise and barrier self-efficacy to engage in leisure-time physical activity during pregnancy. *Ann Behav Med.* 2009;37(3):325-334.
- 39. Williams GC, Grow VM, Freedman ZR, Ryan RM, Deci EL. Motivational predictors of weight loss and weight-loss maintenance. *J Pers Soc Psychol.* 1996;70(1):115-126.
- 40. Silva MN, Markland D, Carraca EV, et al. Exercise autonomous motivation predicts 3-yr weight loss in women. *Med Sci Sports Exerc*. 2011;43(4):728-737.
- 41. Webber KH, Tate DF, Ward DS, Bowling JM. Motivation and its relationship to adherence to self-monitoring and weight loss in a 16-week Internet behavioral weight loss intervention. *J Nutr Educ Behav.* 2010;42(3):161-167.
- 42. Koestner R, Otis N, Powers TA, Pelletier L, Gagnon H. Autonomous motivation, controlled motivation, and goal progress. *J Pers.* 2008;76(5):1201-1230.
- 43. Chang MW, Nitzke S, Brown R. Mothers In Motion intervention effect on psychosocial health in young, low-income women with overweight or obesity. *BMC Public Health*. 2019;19(1):56.
- 44. Chang MW, Brown R, Nitzke S. A Community-Based Intervention Program's Effects on Dietary Intake Behaviors. *Obesity (Silver Spring)*. 2017;25(12):2055-2061.
- 45. Chang M, Brown R, Wegner DT. Perceived Stress Can Mediate the Associations between a Lifestyle Intervention and Fat and Fast Food Intakes. . *The Academic Nutrition and Dietetics* Under review.
- 46. Chang M, Brown R, Wegener DT. Psychosocial Factors Mediated the Association Between Stress and Depressive Symptoms in Low-Income Overweight or Obesity Mother of Young Children. *STress and Health*. Under review.
- 47. Chang M, Robbins L, Ling J, Brown R, Wegener D. Mediators Affecting the Association between Intervention and Stress in Low-Income women with Overweight or Obesity. *Journal of Health Psychology*. 2019.
- 48. Chang M, Shaffir J, Brown R, Wegener D. Mediation by Self-Efficacy in the Relation between Social Support and Dietary Intake in Low-Income Postpartum Women Who were Overweight or Obese. .. doi: 10.1016/j.appet.2019.05.031. Epub 2019 May 26. *Appetite*. 2019

- 49. Chang M, Tan A, Ling J, Wegener DT, Robbins L. Mediators of Intervention Effects on Dietary Fat Intake in Low-Income Overweight or Obese Women With Young Children. *Appetite*. 2020.
- 50. Chang MW, Hales D, Brown R, Ward D, Resnicow K, Nitzke S. Validation of PIN 3 physical activity survey in low-income overweight and obese young mothers. *BMC Public Health*. 2015;15:121.
- 51. Schacter DL, Benoit RG, De Brigard F, Szpunar KK. Episodic future thinking and episodic counterfactual thinking: intersections between memory and decisions. *Neurobiol Learn Mem.* 2015;117:14-21.
- 52. LaCroix AZ, Bellettiere J, Rillamas-Sun E, et al. Association of Light Physical Activity Measured by Accelerometry and Incidence of Coronary Heart Disease and Cardiovascular Disease in Older Women. *JAMA Netw Open.* 2019;2(3):e190419.
- 53. Matthews CE, Keadle SK, Troiano RP, et al. Accelerometer-measured dose-response for physical activity, sedentary time, and mortality in US adults. *Am J Clin Nutr.* 2016;104(5):1424-1432.
- 54. LaMonte MJ, Buchner DM, Rillamas-Sun E, et al. Accelerometer-Measured Physical Activity and Mortality in Women Aged 63 to 99. *J Am Geriatr Soc.* 2018;66(5):886-894.
- 55. LaMonte MJ, Lewis CE, Buchner DM, et al. Both Light Intensity and Moderate-to-Vigorous Physical Activity Measured by Accelerometry Are Favorably Associated With Cardiometabolic Risk Factors in Older Women: The Objective Physical Activity and Cardiovascular Health (OPACH) Study. *J Am Heart Assoc.* 2017;6(10).
- 56. Practice CoO. Exercise during pregnancy and postpartum period. <a href="https://www.acog.org/Clinical-Guidance-and-Publications/Committee-Opinions/Committee-on-Obstetric-Practice/Physical-Activity-and-Exercise-During-Pregnancy-and-the-Postpartum-Period">https://www.acog.org/Clinical-Guidance-and-Publications/Committee-Opinions/Committee-on-Obstetric-Practice/Physical-Activity-and-Exercise-During-Pregnancy-and-the-Postpartum-Period</a>. Published 2017. Accessed August 15, 2018.
- 57. Han TS, van Leer EM, Seidell JC, Lean ME. Waist circumference action levels in the identification of cardiovascular risk factors: prevalence study in a random sample. *BMJ*. 1995;311(7017):1401-1405.
- 58. van Dis I, Kromhout D, Geleijnse JM, Boer JM, Verschuren WM. Body mass index and waist circumference predict both 10-year nonfatal and fatal cardiovascular disease risk: study conducted in 20,000 Dutch men and women aged 20-65 years. *Eur J Cardiovasc Prev Rehabil*. 2009;16(6):729-734.
- 59. Lavie CJ, De Schutter A, Patel D, Artham SM, Milani RV. Body composition and coronary heart disease mortality--an obesity or a lean paradox? *Mayo Clin Proc.* 2011;86(9):857-864.
- 60. Mokdad AH, Ford ES, Bowman BA, et al. Prevalence of obesity, diabetes, and obesity-related health risk factors, 2001. *JAMA*. 2003;289(1):76-79.
- 61. Ryu S, Frith E, Pedisic Z, Kang M, Loprinzi PD. Secular trends in the association between obesity and hypertension among adults in the United States, 1999-2014. *Eur J Intern Med.* 2019;62:37-42.
- 62. Pistoia F, Sacco S, Degan D, Tiseo C, Ornello R, Carolei A. Hypertension and Stroke: Epidemiological Aspects and Clinical Evaluation. *High Blood Press Cardiovasc Prev.* 2016;23(1):9-18.
- 63. Schacter DL, Addis DR, Buckner RL. Remembering the past to imagine the future: the prospective brain. *Nat Rev Neurosci*. 2007;8(9):657-661.
- 64. Stawarczyk D, D'Argembeau A. Neural correlates of personal goal processing during episodic future thinking and mind-wandering: An ALE meta-analysis. *Hum Brain Mapp.* 2015;36:2929-2947.
- 65. Benoit RG, Schacter DL. Specifying the core network supporting episodic simulation and episodic memory by activation likelihood estimation. *Neuropsychologia*. 2015;75:450-457.
- 66. Takeuchi H, Taki Y, Sassa Y, et al. Brain structures associated with executive functions during everyday events in a non-clinical sample. *Brain Struct Funct*. 2013;218(4):1017-1032.
- 67. Schacter DL, Benoit RG, Szpunar KK. Episodic Future Thinking: Mechanisms and Functions. *Curr Opin Behav Sci.* 2017;17:41-50.
- 68. Palombo DJ, Hayes SM, Peterson KM, Keane MM, Verfaellie M. Medial Temporal Lobe Contributions to Episodic Future Thinking: Scene Construction or Future Projection? *Cereb Cortex.* 2018;28(2):447-458.
- 69. Peters J, Buchel C. Episodic future thinking reduces reward delay discounting through an enhancement of prefrontal-mediotemporal interactions. *Neuron*. 2010;66(1):138-148.
- 70. Bandura A. Health promotion by social cognitive means. *Health Educ Behav.* 2004;31(2):143-164.
- 71. Foundation M. Research Network on SES and Health. <a href="https://macses.ucsf.edu/research/psychosocial/socsupp.php">https://macses.ucsf.edu/research/psychosocial/socsupp.php</a>. Published 2008. Accessed April 26, 2020.
- 72. Rebetez MM, Barsics C, Rochat L, D'Argembeau A, Van der Linden M. Procrastination, consideration of future consequences, and episodic future thinking. *Conscious Cogn.* 2016;42:286-292.
- 73. Bandura A. Social learning theory. Englewood Cliffs, N.J.: Prentice-Hall; 1977.
- 74. MacLeod AD. Prospection, well-being and memory *Memory Studies*. 2016;9:266-274.

- 75. Miloyan B, Bulley A, Suddendorf T. Episodic foresight and anxiety: Proximate and ultimate perspectives. *Br J Clin Psychol.* 2016;55(1):4-22.
- 76. Wu JQ, Szpunar KK, Godovich SA, Schacter DL, Hofmann SG. Episodic future thinking in generalized anxiety disorder. *J Anxiety Disord*. 2015;36:1-8.
- 77. Diamond A. Executive functions. *Annu Rev Psychol.* 2013;64:135-168.
- 78. Dohle S, Diel K, Hofmann W. Executive functions and the self-regulation of eating behavior: A review. *Appetite*. 2018;124:4-9.
- 79. Appelhans BM, Waring ME, Schneider KL, et al. Delay discounting and intake of ready-to-eat and away-from-home foods in overweight and obese women. *Appetite*. 2012;59(2):576-584.
- 80. Dassen FC, Jansen A, Nederkoorn C, Houben K. Focus on the future: Episodic future thinking reduces discount rate and snacking. *Appetite*. 2016;96:327-332.
- 81. Stein JS, Sze YY, Athamneh L, Koffarnus MN, Epstein LH, Bickel WK. Think fast: rapid assessment of the effects of episodic future thinking on delay discounting in overweight/obese participants. *J Behav Med*. 2017;40(5):832-838.
- 82. Vartanian LR, Chen WH, Reily NM, Castel AD. The parallel impact of episodic memory and episodic future thinking on food intake. *Appetite*. 2016;101:31-36.
- 83. Sze YY, Daniel TO, Kilanowski CK, Collins RL, Epstein LH. Web-Based and Mobile Delivery of an Episodic Future Thinking Intervention for Overweight and Obese Families: A Feasibility Study. *JMIR Mhealth Uhealth*. 2015;3(4):e97.
- 84. Lin H, Epstein LH. Living in the moment: effects of time perspective and emotional valence of episodic thinking on delay discounting. *Behav Neurosci.* 2014;128(1):12-19.
- 85. D'Argembeau A, Stawarczyk D, Majerus S, et al. The neural basis of personal goal processing when envisioning future events. *J Cogn Neurosci*. 2010;22(8):1701-1713.
- 86. McFarland CP, Primosch M, Maxson CM, Stewart BT. Enhancing memory and imagination improves problem solving among individuals with depression. *Mem Cognit*. 2017;45(6):932-939.
- 87. Terrett G, Rose NS, Henry JD, et al. The relationship between prospective memory and episodic future thinking in younger and older adulthood. *Q J Exp Psychol (Hove)*. 2016;69(2):310-323.
- 88. Schacter DL. Adaptive constructive processes and the future of memory. *Am Psychol.* 2012;67(8):603-613.
- 89. Thorstad R, Wolff P. A big data analysis of the relationship between future thinking and decision-making. *Proc Natl Acad Sci U S A.* 2018;115(8):E1740-E1748.
- 90. Bandura A. The Primacy of Self-Regulation in Health Promotion. *Applied Psychology*. 2005;54(2):245-254.
- 91. Huang Y, Lv W, Wu J. Relationship Between Intrinsic Motivation and Undergraduate Students' Depression and Stress: The Moderating Effect of Interpersonal Conflict. *Psychol Rep.* 2016;119(2):527-538.
- 92. Barch DM, Yodkovik N, Sypher-Locke H, Hanewinkel M. Intrinsic motivation in schizophrenia: relationships to cognitive function, depression, anxiety, and personality. *J Abnorm Psychol.* 2008;117(4):776-787.
- 93. Brown AD, Kouri NA, Rahman N, Joscelyne A, Bryant RA, Marmar CR. Enhancing self-efficacy improves episodic future thinking and social-decision making in combat veterans with posttraumatic stress disorder. *Psychiatry Res.* 2016:242:19-25.
- 94. Young MD, Plotnikoff RC, Collins CE, Callister R, Morgan PJ. Social cognitive theory and physical activity: a systematic review and meta-analysis. *Obes Rev.* 2014;15(12):983-995.
- 95. Simons J, Vansteenkiste M, Lens W. Placing Motivation and Future Time Perspective Theory in a Temporal Perspective. *Educational Psychology Review*. 2004;16(2):121-139.
- 96. Santos I, Mata J, Silva MN, Sardinha LB, Teixeira PJ. Predicting long-term weight loss maintenance in previously overweight women: a signal detection approach. *Obesity (Silver Spring)*. 2015;23(5):957-964.
- 97. Teixeira PJ, Silva MN, Mata J, Palmeira AL, Markland D. Motivation, self-determination, and long-term weight control. *Int J Behav Nutr Phys Act.* 2012;9:22.
- 98. Izard C. The Many Meanings/Aspects of Emotion: Definitions, Functions, Activation, and Regulation. *Emotion Review* 2010;2(4):363-370.
- 99. Muraven M, Baumeister RF. Self-regulation and depletion of limited resources: does self-control resemble a muscle? *Psychol Bull.* 2000;126(2):247-259.
- 100. Diamond A, Ling DS. Conclusions about interventions, programs, and approaches for improving executive functions that appear justified and those that, despite much hype, do not. *Dev Cogn Neurosci.* 2016;18:34-48.

- 101. Best JR, Nagamatsu LS, Liu-Ambrose T. Improvements to executive function during exercise training predict maintenance of physical activity over the following year. *Front Hum Neurosci.* 2014;8:353.
- 102. Emery RL, Levine MD. Questionnaire and behavioral task measures of impulsivity are differentially associated with body mass index: A comprehensive meta-analysis. *Psychol Bull.* 2017;143(8):868-902.
- 103. Yang Y, Shields GS, Guo C, Liu Y. Executive function performance in obesity and overweight individuals: A meta-analysis and review. *Neurosci Biobehav Rev.* 2018;84:225-244.
- Wu M, Brockmeyer T, Hartmann M, Skunde M, Herzog W, Friederich HC. Set-shifting ability across the spectrum of eating disorders and in overweight and obesity: a systematic review and meta-analysis. *Psychol Med.* 2014;44(16):3365-3385.
- 105. Weller RE, Cook EW, 3rd, Avsar KB, Cox JE. Obese women show greater delay discounting than healthy-weight women. *Appetite*. 2008;51(3):563-569.
- 106. Christian BM, Miles LK, Fung FH, Best S, Macrae CN. The shape of things to come: exploring goal-directed prospection. *Conscious Cogn.* 2013;22(2):471-478.
- 107. D'Argembeau A. Reasoning as memory. In: Feeney A, Thompson VA, eds. *Knolwedge structures involved in episodic future thinking*. Hove, UK: Psychology Press; 2015:128–145.
- 108. Fishbach A, Ferguson MJ. Social psychology: The goal construct in social psychology. In: Kruglanski AW, Higgins ET, eds. *Handbook of basic principles*. 2nd ed. New York: Guilford Press; 2007:490–515.
- 109. Szpunar KK, Spreng N, Schacter DL. A taxonomy of prospection: Introducing an organizational framework for future-oriented cognition. *PNAS*. 2014;111(52):18414-18421.
- 110. Reeve J, Ryan R, Deci EL, Jang H. Understanding and promoting autonomous self-regulation: A self-determination theory perspective. In: Schunk DH, Zimmerman BJ, eds. *Motivation and self-regulated learning: Theory, research, and applications.* Lawrence Erlbaum Associates Publishers; 2008:223–244.
- 111. Aronson E. The power of self-persuasion. *American Psychologist*. 1999;54(11):875–884.
- 112. Institute NC. Percentage energy from fat short instrument (PFat). <a href="http://appliedresearch.cancer.gov/diet/screeners/fat/">http://appliedresearch.cancer.gov/diet/screeners/fat/</a>. Published 1996. Accessed January 1, 2018.
- 113. Institute NC. Five-factor screener: National Health Interview Survey (NHIS) diet and nutrition. 2005.
- 114. Institute NC. Five-factor screener: National Health Interview Survey (NHIS) validation results. <a href="https://www.phenxtoolkit.org/index.php?pageLink=browse.si.additionalinfo&id=50000">https://www.phenxtoolkit.org/index.php?pageLink=browse.si.additionalinfo&id=50000</a>. Published 2005. Accessed January 1, 2018.
- 115. Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. *Int J Behav Nutr Phys Act.* 2011;8:115.
- Pelletier LG, Tuson KM, Haddad NK. Client Motivation for Therapy Scale: a measure of intrinsic motivation, extrinsic motivation, and amotivation for therapy. *J Pers Assess.* 1997;68(2):414-435.
- 117. Luszczynska A, Scholz U, Schwarzer R. The general self-efficacy scale: multicultural validation studies. *J Psychol.* 2005;139(5):439-457.
- 118. Chang M, Nitzke S, Brown R, Baumann L, Oakley L. Development and validation of a self-efficacy measure for fat intake behaviors in low-income women. *J Nutr Educ Behav.* 2003;35(6):302-307.
- 119. Chang M, Brown R, Nitzke S. Scale development: Factors affecting diet, exercise, and stress management (FADESM). *BMC Public Health*. 2008;8(76).
- 120. Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. *J Pers Soc Psychol*. 2003;85(2):348-362.
- 121. Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. *J Health Soc Behav.* 1983;24(4):385-396.
- 122. Barratt ES. Anxiety and impulsiveness related to psychomotor efficiency. *Perceptual and Motor Skills*. 1959;9:191–198.
- 123. Chang MW, Nitzke S, Buist D, Cain D, Horning S, Eghtedary K. I am pregnant and want to do better but i can't: focus groups with low-income overweight and obese pregnant women. *Matern Child Health J.* 2015;19(5):1060-1070.
- 124. Chang MW, Brown R, Nitzke S. Results and lessons learned from a prevention of weight gain program for low-income overweight and obese young mothers: Mothers In Motion. *BMC Public Health*. 2017;17(1):182.
- 125. Gollwitzer PM. Implementation intentions: Strong effects of simple plans. *American Psychologist*. 1999;54(7):493-503.

Adams C, Rennie L, Uskul AK, Appleton KM. Visualising future behaviour: Effects for snacking on biscuit bars,

126.